CLINICAL TRIAL: NCT01884233
Title: Cell Phone Technology Targeting ART Adherence and Drug Use
Acronym: TXT-CBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Suzette Glasner-Edwards, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R34DA033196 (NIH); 1R34DA033196 (NIH)
Record Dates: First submitted 2013-05-24; First posted 2013-06-21 (Estimated); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: HIV; Opioid Abuse
Keywords: HIV; Opioid Abuse; Mobile technology
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Text Messaging CBT (TXT-CBT) (Experimental): This condition will receive CBT based text messaging (TXT-CBT). Those assigned to TXT-CBT will also be given a treatment manual (developed in Phase I) containing descriptions of core therapeutic content/topics for each week. HIV-infected participants will have an initial meeting with a CBT clinician to review the Life-Steps concepts. The 3 most applicable medication adherence skills will be identified for emphasis in tailored messages. A research coordinator will meet with the participants weekly at data collection visits throughout the intervention phase to answer any technical questions and ensure that the intervention program is working properly.
  Interventions: Behavioral: Standard Care; Behavioral: Text Messaging CBT (TXT-CBT)
- Standard Care (Active Comparator): Those assigned to the Standard Care condition will receive the standard monthly medical management physician visit typically associated with HIV care. In addition, a pamphlet with information about HIV, the importance of ART adherence, and relapse prevention will be provided to participants in this condition.
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Standard Care — Standard care will include usual treatment for HIV and a pamphlet that will be provided to the participants with information about ART adherence and relapse prevention.
Behavioral: Text Messaging CBT (TXT-CBT) — Those assigned to TXT-CBT will be given a treatment manual (developed in Phase I) containing descriptions of core therapeutic content/topics for each week. HIV-infected participants will have initial meeting with a CBT clinician to review the core CBT concepts for promoting ART adherence. The 3 most applicable medication adherence skills will be identified for emphasis in tailored messages. A research coordinator will meet with the participants weekly at data collection visits throughout the intervention phase to answer any technical questions and ensure that the intervention program is working properly.
  Arms: Text Messaging CBT (TXT-CBT)

SUMMARY:
The objective of the current research is to improve treatment for injection opioid users by augmenting pharmacotherapy with an innovative text-messaging strategy to promote relapse prevention skills, reduce HIV-risk behaviors, and improve HIV treatment regimen adherence.

DETAILED DESCRIPTION:
the specific aims of this research are 1) To develop and refine, with user feedback, a cognitive behavioral therapy-based text-messaging intervention (TXT-CBT) for HIV-infected adults with opioid dependence; 2) To conduct a pilot randomized clinical trial to assess the feasibility of recruiting and retaining individuals for a large scale study and to determine the effect size of TXT-CBT over and above standard care (SC) on opioid use, HIV medication adherence, and healthcare outcomes. Both SC and SC+TXT-CBT participants will be assessed at baseline, treatment-end, and 12 weeks post-treatment; and 3) To examine potential mechanisms of action of TXT-CBT, including self-efficacy, affect regulation, and social support. The investigators hypothesize that TXT-CBT delivered in conjunction with SC will produce greater reductions in opioid use and HIV-risk behaviors, and will improve HIV treatment regimen adherence, relative to MM alone. Further, the investigators expect that SC+TXT-CBT will facilitate greater changes in negative affect, self-efficacy, and social support, and these changes will be associated with substance use outcomes. TXT-CBT incorporates specific substance- and adherence-focused cognitive therapy techniques with a concurrent emphasis on reducing HIV-risk behaviors. By providing support to maximize HIV treatment regimen adherence, coupled with coping skills to address withdrawal symptoms and stress, two important factors in opioid relapse, TXT-CBT may provide a promising, cost-effective, and easily deployable augmenting strategy for the treatment of opioid users who are HIV-infected.

ELIGIBILITY:
Inclusion criteria for participants in both Phase I and Phase II will be:

1. Age 18 or older;
2. DSM-IV diagnosis of Opioid Dependence;
3. HIV-infected serostatus;
4. Able to provide informed consent;
5. Willing and able to participate in study procedures,
6. Good general health or, in the case of a medical/psychiatric condition needing ongoing treatment, potential participant should be under the care of a physician who provides documented willingness to continue participant's medical management and coordinate care with the study physicians.

Exclusion Criteria:

1. Lack of proficiency in English;
2. Currently homeless (unless residing in a recovery home for which contact information can be provided);
3. Dependence on an illicit substance for which medical detoxification is imminently needed.
4. Presence of clinically significant psychiatric symptoms as assessed by MINI, such as psychosis, acute mania, or suicide risk that would require immediate treatment or make study compliance difficult.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2012-12; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in Substance Use | The ASI is to be collected at baseline (week 0), treatment-end (week 12), and Follow-Up (wek 24). UDS is collected weekly during the intervetion.
  Addiction Severity Index (ASI) is an instrument widely used in addiction research to quantify drug use frequency and related problem areas. Urine Drug Screen (UDS). Urine drug screens will be collected monthly using temperature controlled test cups. An FDA-approved one-step test will be used. During the 12-week treatment period, one full-screen panel and two panels only testing for opioids (heroin and prescription opioids) will be conducted. The UDS will test for the presence of: amphetamines, benzodiazepines, methadone, cocaine, methamphetamine, morphine (heroin), hydrocodone (Vicodin), oxycodone (OxyContin), and marijuana. The participants' change in substance use over time (as assessed by the ASI and UDS results) is being assessed from each timepoint to the next.
Change in HIV Risk Behaviors | RBS will be collected at baseline (week 0), treatment-end (week 12), and FU (week 24)
  Risk Behavior Survey (RBS): The RBS (Darke et al., 1991) is a brief interview assessing involvement in HIV risk behaviors in the areas of drug use and sex in the previous 30 days. Additional items include whether the sexual partner uses or injects drugs. The participants' change in RBS scores is being assessed from each timepoint to the next.
Change in treatment adherence | Pill bottle collection will be weekly during the intervention. Pill counts and Viral load will be collected at baseline (week 0), treatment end (week 12), and FU (week 24).
  ART Adherence. The investigator will use monthly phone-based unannounced pill counts (UPCs); Pharmacy information from pill bottles will also be collected to verify the number of pills dispensed between calls. Self-reported adherence will be assessed monthly using a brief adherence survey developed by Lu et al. Viral load will serve as a biological indicator of adherence. Consistent with the typical frequency with which viral load is assessed in clinical settings, data concerning viral load will be collected at baseline (week 0), treatment end (week 12), and FU (week 24) via chart review from the participant's medical provider. The participants' change in Adherence scores is being assessed from each timepoint to the next.

SECONDARY OUTCOMES:
Change in health-related quality of life | week 0, week 12 and week 24
  Data concerning health-related quality of life during and after treatment will be collected using the SF-12 Health Survey that uses just 12 questions to measure functional health and well-being from the patient's point of view

CONTACTS AND LOCATIONS:
Overall Officials: Suzette Glasner, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Isap Ocrc, Los Angeles, California, United States